CLINICAL TRIAL: NCT02762851
Title: A Randomized Controlled Trial of Influenza Vaccine to Prevent Adverse Vascular Events
Brief Title: Influenza Vaccine To Prevent Adverse Vascular Events (RCT-IVVE)
Acronym: RCT-IVVE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RCT-IVVE 2015
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Heart Failure; Influenza
Keywords: Influenza; Vaccine; Heart failure; Vascular
MeSH Terms: conditions — Heart Failure; Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Influenza vaccine (Experimental): Participants at high risk for adverse vascular events will be immunized with 0.5 ml dose of inactivated trivalent influenza vaccine prior to the influenza season.
  Interventions: Drug: inactivated trivalent influenza vaccine
- Placebo vaccine (Placebo Comparator): Participants at high risk for adverse vascular events will be vaccinated with a 0.5 ml dose of sterile saline prior to the influenza season.
  Interventions: Other: Sterile saline

INTERVENTIONS:
Other: Sterile saline — 0.5 ml dose injected intramuscularly
  Arms: Placebo vaccine
Drug: inactivated trivalent influenza vaccine — 0.5 ml dose injected intramuscularly
  Other Names: VAXIGRIP vaccine
  Arms: Influenza vaccine

SUMMARY:
A multi-centre, randomized, placebo controlled, trial. Participants at high-risk for vascular events from the network of INTER- CHF will be randomized to inactivated influenza vaccine or placebo and followed prospectively over three influenza seasons. 5,000 participants will be enrolled prior to influenza season, randomized to either influenza vaccine or saline placebo, either of which they will receive annually for three years and then followed over each of the influenza seasons.

DETAILED DESCRIPTION:
Cardiovascular disease is a major cause of morbidity and mortality. There is recent evidence that infection due to influenza may precipitate vascular events such as myocardial infarctions and strokes. There is some evidence that influenza vaccination may prevent such events but the data are inconclusive. The investigators propose a randomized controlled trial to assess whether influenza vaccination will prevent vascular illness. Adults with clinical heart failure will be randomized to inactivated influenza vaccine or saline placebo each year for three consecutive years. They will be followed over six months for a composite of cardiovascular death, non-fatal myocardial infarction, non-fatal stroke and hospitalizations for heart failure using standardized criteria. Rigorous demonstration of influenza vaccine leading to a reduction in major adverse vascular events in patients with heart failure would lead to a major change in how these patients are managed. Given the large burden of disease both in Canada and globally, the possibility to reduce cardiovascular and stroke related death is a compelling reason to conduct this trial.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and NYHA (New York Heart Association) functional class II, III and IV

Exclusion Criteria:

* Anaphylactic reaction to a previous dose of TIV(trivalent influenza vaccine)
* Known IgE( Immunoglobulin E)-mediated hypersensitivity to eggs manifested as hives, swelling of the mouth and throat, difficulty in breathing, hypotension, or shock
* Guillain-Barré syndrome within eight weeks of a previous influenza vaccine
* Anaphylactic reaction to neomycin
* Patients who have had influenza vaccine in two of the three previous years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Adverse cardiovascular event | Six months
  The primary outcome will be a composite of cardiovascular death, non-fatal myocardial infarction, non-fatal stroke and hospitalizations for heart failure using standardized criteria.

SECONDARY OUTCOMES:
Cardiovascular (CV) death | Six months
  CV death alone will be a secondary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Loeb, MD, MSc., Principal Investigator — McMaster University
Locations (13):
- Douala General Hospital, Douala, Cameroon
- Fuwai Hospital, Beijing, Xicheng District, China
- Centre for Chronic Disease Control, New Delhi, India
- Aga Khan University, Nairobi, Kenya
- American University of Beirut Medical Center, Beirut, Lebanon
- Maputo Central Hospital (Full Trial), Maputo, Mozambique
- Bayero University and Aminu Kano Teaching Hospital, Kano, Nigeria
- University of Philippines, Manila, Emita, Philippines
- King Saud Univeristy, Riyadh, Saudi Arabia
- AlShaab Teaching Hospital, Khartoum, Sudan
- Mulago Hospital, Kampala, Uganda
- Sheikh Khalifa Medical City, Abu Dhabi, United Arab Emirates
- University of Zambia School of Medicine, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Causes of death 2008, World Health Organization, Geneva, http://www.who.int/healthinfo/ global_burden_disease/ cod_2008_sources_methods.pdf.
- [Background] Statistics Canada. Morality, Summary List of Causes 2008. Released October 18, 2011.
- [Background] Tracking Heart Disease and Stroke in Canada. Released June 2009
- [Background] Remme WJ, Torp-Pedersen C, Cleland JG, Poole-Wilson PA, Metra M, Komajda M, Swedberg K, Di Lenarda A, Spark P, Scherhag A, Moullet C, Lukas MA. Carvedilol protects better against vascular events than metoprolol in heart failure: results from COMET. J Am Coll Cardiol. 2007 Mar 6;49(9):963-71. doi: 10.1016/j.jacc.2006.10.059. Epub 2007 Feb 20. PMID 17336720
- [Background] Gheorghiade M, Bohm M, Greene SJ, Fonarow GC, Lewis EF, Zannad F, Solomon SD, Baschiera F, Botha J, Hua TA, Gimpelewicz CR, Jaumont X, Lesogor A, Maggioni AP; ASTRONAUT Investigators and Coordinators. Effect of aliskiren on postdischarge mortality and heart failure readmissions among patients hospitalized for heart failure: the ASTRONAUT randomized trial. JAMA. 2013 Mar 20;309(11):1125-35. doi: 10.1001/jama.2013.1954. PMID 23478743
- [Background] Massie BM, Carson PE, McMurray JJ, Komajda M, McKelvie R, Zile MR, Anderson S, Donovan M, Iverson E, Staiger C, Ptaszynska A; I-PRESERVE Investigators. Irbesartan in patients with heart failure and preserved ejection fraction. N Engl J Med. 2008 Dec 4;359(23):2456-67. doi: 10.1056/NEJMoa0805450. Epub 2008 Nov 11. PMID 19001508
- [Background] Bohm M, Swedberg K, Komajda M, Borer JS, Ford I, Dubost-Brama A, Lerebours G, Tavazzi L; SHIFT Investigators. Heart rate as a risk factor in chronic heart failure (SHIFT): the association between heart rate and outcomes in a randomised placebo-controlled trial. Lancet. 2010 Sep 11;376(9744):886-94. doi: 10.1016/S0140-6736(10)61259-7. PMID 20801495
- [Background] Homma S, Thompson JL, Pullicino PM, Levin B, Freudenberger RS, Teerlink JR, Ammon SE, Graham S, Sacco RL, Mann DL, Mohr JP, Massie BM, Labovitz AJ, Anker SD, Lok DJ, Ponikowski P, Estol CJ, Lip GY, Di Tullio MR, Sanford AR, Mejia V, Gabriel AP, del Valle ML, Buchsbaum R; WARCEF Investigators. Warfarin and aspirin in patients with heart failure and sinus rhythm. N Engl J Med. 2012 May 17;366(20):1859-69. doi: 10.1056/NEJMoa1202299. Epub 2012 May 2. PMID 22551105
- [Background] Kinlay S, Ganz P. Role of endothelial dysfunction in coronary artery disease and implications for therapy. Am J Cardiol. 1997 Nov 6;80(9A):11I-16I. doi: 10.1016/s0002-9149(97)00793-5. PMID 9375937
- [Background] Chan NN, Colhoun HM, Vallance P. Cardiovascular risk factors as determinants of endothelium-dependent and endothelium-independent vascular reactivity in the general population. J Am Coll Cardiol. 2001 Dec;38(7):1814-20. doi: 10.1016/s0735-1097(01)01669-2. PMID 11738279
- [Background] Davies MJ. The composition of coronary-artery plaques. N Engl J Med. 1997 May 1;336(18):1312-4. doi: 10.1056/NEJM199705013361809. No abstract available. PMID 9113937
- [Background] Wanishsawad C, Zhou YF, Epstein SE. Chlamydia pneumoniae-induced transactivation of the major immediate early promoter of cytomegalovirus: potential synergy of infectious agents in the pathogenesis of atherosclerosis. J Infect Dis. 2000 Feb;181(2):787-90. doi: 10.1086/315235. PMID 10669378
- [Background] Conti CR. Vascular events responsible for thrombotic occlusion of a blood vessel. Clin Cardiol. 1993 Nov;16(11):761-2. doi: 10.1002/clc.4960161103. PMID 8269651
- [Background] Lundman P, Eriksson M, Schenck-Gustafsson K, Karpe F, Tornvall P. Transient triglyceridemia decreases vascular reactivity in young, healthy men without risk factors for coronary heart disease. Circulation. 1997 Nov 18;96(10):3266-8. doi: 10.1161/01.cir.96.10.3266. PMID 9396413
- [Background] Kawano H, Motoyama T, Hirashima O, Hirai N, Miyao Y, Sakamoto T, Kugiyama K, Ogawa H, Yasue H. Hyperglycemia rapidly suppresses flow-mediated endothelium-dependent vasodilation of brachial artery. J Am Coll Cardiol. 1999 Jul;34(1):146-54. doi: 10.1016/s0735-1097(99)00168-0. PMID 10400004
- [Background] Gwini SM, Coupland CA, Siriwardena AN. The effect of influenza vaccination on risk of acute myocardial infarction: self-controlled case-series study. Vaccine. 2011 Feb 1;29(6):1145-9. doi: 10.1016/j.vaccine.2010.12.017. Epub 2010 Dec 18. PMID 21172383
- [Background] Naghavi M, Barlas Z, Siadaty S, Naguib S, Madjid M, Casscells W. Association of influenza vaccination and reduced risk of recurrent myocardial infarction. Circulation. 2000 Dec 19;102(25):3039-45. doi: 10.1161/01.cir.102.25.3039. PMID 11120692
- [Background] Meyers D, Beahm D, Jurisich P, Milford C, Edlavich S. Influenza and pneumococcal vaccinations fail to prevent myocardial infarction. Heart Drug. 2004;4:96 -100.
- [Background] Lavallee P, Perchaud V, Gautier-Bertrand M, Grabli D, Amarenco P. Association between influenza vaccination and reduced risk of brain infarction. Stroke. 2002 Feb;33(2):513-8. doi: 10.1161/hs0202.102328. PMID 11823662
- [Background] Siscovick DS, Raghunathan TE, Lin D, Weinmann S, Arbogast P, Lemaitre RN, Psaty BM, Alexander R, Cobb LA. Influenza vaccination and the risk of primary cardiac arrest. Am J Epidemiol. 2000 Oct 1;152(7):674-7. doi: 10.1093/aje/152.7.674. PMID 11032163
- [Background] Siriwardena AN, Gwini SM, Coupland CA. Influenza vaccination, pneumococcal vaccination and risk of acute myocardial infarction: matched case-control study. CMAJ. 2010 Oct 19;182(15):1617-23. doi: 10.1503/cmaj.091891. Epub 2010 Sep 20. PMID 20855479
- [Background] Heffelfinger JD, Heckbert SR, Psaty BM, Weiss NS, Thompson WW, Bridges CB, Jackson LA. Influenza vaccination and risk of incident myocardial infarction. Hum Vaccin. 2006 Jul-Aug;2(4):161-6. doi: 10.4161/hv.2.4.2943. Epub 2006 Jul 24. PMID 17012887
- [Background] Nichol KL, Nordin J, Mullooly J, Lask R, Fillbrandt K, Iwane M. Influenza vaccination and reduction in hospitalizations for cardiac disease and stroke among the elderly. N Engl J Med. 2003 Apr 3;348(14):1322-32. doi: 10.1056/NEJMoa025028. PMID 12672859
- [Background] Jackson LA, Yu O, Heckbert SR, Psaty BM, Malais D, Barlow WE, Thompson WW; Vaccine Safety Datalink Study Group. Influenza vaccination is not associated with a reduction in the risk of recurrent coronary events. Am J Epidemiol. 2002 Oct 1;156(7):634-40. doi: 10.1093/aje/kwf073. PMID 12244032
- [Background] Armstrong BG, Mangtani P, Fletcher A, Kovats S, McMichael A, Pattenden S, Wilkinson P. Effect of influenza vaccination on excess deaths occurring during periods of high circulation of influenza: cohort study in elderly people. BMJ. 2004 Sep 18;329(7467):660. doi: 10.1136/bmj.38198.594109.AE. Epub 2004 Aug 15. PMID 15313884
- [Background] Wang CS, Wang ST, Lai CT, Lin LJ, Chou P. Impact of influenza vaccination on major cause-specific mortality. Vaccine. 2007 Jan 26;25(7):1196-203. doi: 10.1016/j.vaccine.2006.10.015. Epub 2006 Oct 25. PMID 17097773
- [Background] Johnstone J, Loeb M, Teo KK, Gao P, Dyal L, Liu L, Avezum A, Cardona-Munoz E, Sleight P, Fagard R, Yusuf S; Ongoing Telmisartan Alone and in Combination With Ramipril Global EndPoint Trial (ONTARGET); Telmisartan Randomized Assessment Study in ACE Intolerant Subjects With Cardiovascular Disease (TRANSCEND) Investigators. Influenza vaccination and major adverse vascular events in high-risk patients. Circulation. 2012 Jul 17;126(3):278-86. doi: 10.1161/CIRCULATIONAHA.111.071100. Epub 2012 Jun 19. PMID 22715472
- [Background] Keller T, Weeda VB, van Dongen CJ, Levi M. Influenza vaccines for preventing coronary heart disease. Cochrane Database Syst Rev. 2008 Jul 16;(3):CD005050. doi: 10.1002/14651858.CD005050.pub2. PMID 18646119
- [Background] Warren-Gash C, Smeeth L, Hayward AC. Influenza as a trigger for acute myocardial infarction or death from cardiovascular disease: a systematic review. Lancet Infect Dis. 2009 Oct;9(10):601-10. doi: 10.1016/S1473-3099(09)70233-6. PMID 19778762
- [Background] Udell JA, Zawi R, Bhatt DL, Keshtkar-Jahromi M, Gaughran F, Phrommintikul A, Ciszewski A, Vakili H, Hoffman EB, Farkouh ME, Cannon CP. Association between influenza vaccination and cardiovascular outcomes in high-risk patients: a meta-analysis. JAMA. 2013 Oct 23;310(16):1711-20. doi: 10.1001/jama.2013.279206. PMID 24150467
- [Background] Phrommintikul A, Kuanprasert S, Wongcharoen W, Kanjanavanit R, Chaiwarith R, Sukonthasarn A. Influenza vaccination reduces cardiovascular events in patients with acute coronary syndrome. Eur Heart J. 2011 Jul;32(14):1730-5. doi: 10.1093/eurheartj/ehr004. Epub 2011 Feb 2. PMID 21289042
- [Background] Natarajan P, Cannon CP. Myocardial infarction vaccine? Evidence supporting the influenza vaccine for secondary prevention. Eur Heart J. 2011 Jul;32(14):1701-3. doi: 10.1093/eurheartj/ehr053. Epub 2011 Mar 15. No abstract available. PMID 21406438
- [Background] Canadian Communicable Disease Report 2012. Statement on seasonal influenza vaccine for 2012-2013; 38: 2012.
- [Background] Centers for Disease Control and Prevention (CDC). Prevention and control of influenza with vaccines: recommendations of the Advisory Committee on Immunization Practices (ACIP)--United States, 2012-13 influenza season. MMWR Morb Mortal Wkly Rep. 2012 Aug 17;61(32):613-8. PMID 22895385
- [Background] Blank PR, Schwenkglenks M, Szucs TD. Disparities in influenza vaccination coverage rates by target group in five European countries: trends over seven consecutive seasons. Infection. 2009 Oct;37(5):390-400. doi: 10.1007/s15010-009-8467-y. Epub 2009 Sep 18. PMID 19768382
- [Background] Mereckiene J, Cotter S, Nicoll A, Levy-Bruhl D, Ferro A, Tridente G, Zanoni G, Berra P, Salmaso S, O'Flanagan D, O Flanagan D; VENICE Project Gatekeepers Group. National seasonal influenza vaccination survey in Europe, 2008. Euro Surveill. 2008 Oct 23;13(43):19017. doi: 10.2807/ese.13.43.19017-en. PMID 18947524
- [Background] Population Health Research Institute http://www.phri.ca/
- [Background] ORIGIN Trial Investigators; Gerstein HC, Bosch J, Dagenais GR, Diaz R, Jung H, Maggioni AP, Pogue J, Probstfield J, Ramachandran A, Riddle MC, Ryden LE, Yusuf S. Basal insulin and cardiovascular and other outcomes in dysglycemia. N Engl J Med. 2012 Jul 26;367(4):319-28. doi: 10.1056/NEJMoa1203858. Epub 2012 Jun 11. PMID 22686416
- [Background] ORIGIN Trial Investigators; Bosch J, Gerstein HC, Dagenais GR, Diaz R, Dyal L, Jung H, Maggiono AP, Probstfield J, Ramachandran A, Riddle MC, Ryden LE, Yusuf S. n-3 fatty acids and cardiovascular outcomes in patients with dysglycemia. N Engl J Med. 2012 Jul 26;367(4):309-18. doi: 10.1056/NEJMoa1203859. Epub 2012 Jun 11. PMID 22686415
- [Background] ACCORD Study Group; Gerstein HC, Miller ME, Genuth S, Ismail-Beigi F, Buse JB, Goff DC Jr, Probstfield JL, Cushman WC, Ginsberg HN, Bigger JT, Grimm RH Jr, Byington RP, Rosenberg YD, Friedewald WT. Long-term effects of intensive glucose lowering on cardiovascular outcomes. N Engl J Med. 2011 Mar 3;364(9):818-28. doi: 10.1056/NEJMoa1006524. PMID 21366473
- [Background] CURRENT-OASIS 7 Investigators; Mehta SR, Bassand JP, Chrolavicius S, Diaz R, Eikelboom JW, Fox KA, Granger CB, Jolly S, Joyner CD, Rupprecht HJ, Widimsky P, Afzal R, Pogue J, Yusuf S. Dose comparisons of clopidogrel and aspirin in acute coronary syndromes. N Engl J Med. 2010 Sep 2;363(10):930-42. doi: 10.1056/NEJMoa0909475. PMID 20818903
- [Background] ACCORD Study Group; Ginsberg HN, Elam MB, Lovato LC, Crouse JR 3rd, Leiter LA, Linz P, Friedewald WT, Buse JB, Gerstein HC, Probstfield J, Grimm RH, Ismail-Beigi F, Bigger JT, Goff DC Jr, Cushman WC, Simons-Morton DG, Byington RP. Effects of combination lipid therapy in type 2 diabetes mellitus. N Engl J Med. 2010 Apr 29;362(17):1563-74. doi: 10.1056/NEJMoa1001282. Epub 2010 Mar 14. PMID 20228404
- [Background] ACCORD Study Group; Cushman WC, Evans GW, Byington RP, Goff DC Jr, Grimm RH Jr, Cutler JA, Simons-Morton DG, Basile JN, Corson MA, Probstfield JL, Katz L, Peterson KA, Friedewald WT, Buse JB, Bigger JT, Gerstein HC, Ismail-Beigi F. Effects of intensive blood-pressure control in type 2 diabetes mellitus. N Engl J Med. 2010 Apr 29;362(17):1575-85. doi: 10.1056/NEJMoa1001286. Epub 2010 Mar 14. PMID 20228401
- [Background] Action to Control Cardiovascular Risk in Diabetes Study Group; Gerstein HC, Miller ME, Byington RP, Goff DC Jr, Bigger JT, Buse JB, Cushman WC, Genuth S, Ismail-Beigi F, Grimm RH Jr, Probstfield JL, Simons-Morton DG, Friedewald WT. Effects of intensive glucose lowering in type 2 diabetes. N Engl J Med. 2008 Jun 12;358(24):2545-59. doi: 10.1056/NEJMoa0802743. Epub 2008 Jun 6. PMID 18539917
- [Background] DataFax - Data Management Software for Clinical Trials. http://www.datafax.com/; accessed February 15, 2013.
- [Derived] Loeb M, Roy A, Dokainish H, Dans A, Palileo-Villanueva LM, Karaye K, Zhu J, Liang Y, Goma F, Damasceno A, Alhabib KF, Yonga G, Mondo C, Almahmeed W, Al Mulla A, Thanabalan V, Rao-Melacini P, Grinvalds A, McCready T, Bangdiwala SI, Yusuf S; Influenza Vaccine to Prevent Adverse Vascular Events investigators. Influenza vaccine to reduce adverse vascular events in patients with heart failure: a multinational randomised, double-blind, placebo-controlled trial. Lancet Glob Health. 2022 Dec;10(12):e1835-e1844. doi: 10.1016/S2214-109X(22)00432-6. PMID 36400089
- [Derived] Loeb M, Dokainish H, Dans A, Palileo-Villanueva LM, Roy A, Karaye K, Zhu J, Liang Y, Goma F, Damasceno A, AlHabib KF, Yonga G, Mondo C, Almahmeed W, Al Mulla A, Yusuf S; IVVE investigators. Randomized controlled trial of influenza vaccine in patients with heart failure to reduce adverse vascular events (IVVE): Rationale and design. Am Heart J. 2019 Jun;212:36-44. doi: 10.1016/j.ahj.2019.02.009. Epub 2019 Mar 11. PMID 30933856